CLINICAL TRIAL: NCT00002207
Title: A Randomized, Double-Blind Study of the Antiviral Activity of Once-Daily and Twice-Daily Dosing of Didanosine in Combination With Twice-Daily Dosing of Stavudine in HIV-Infected Subjects
Brief Title: A Comparison of Two Dose Levels of Didanosine Used in Combination With Stavudine in HIV-Infected Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 039D; AI454-143
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2011-04-25 (Estimated); Status verified 2011-04

CONDITIONS: HIV Infections
Keywords: Didanosine; Drug Therapy, Combination; Stavudine; Reverse Transcriptase Inhibitors
MeSH Terms: conditions — HIV Infections | interventions — Stavudine; Didanosine

INTERVENTIONS:
Drug: Stavudine
Drug: Didanosine

SUMMARY:
The purpose of this study is to compare the effectiveness of taking didanosine (ddI) once a day plus stavudine (d4T) twice a day with taking ddI twice a day plus d4T twice a day. This study also examines the safety of giving ddI with d4T in the short-term.

DETAILED DESCRIPTION:
Patients are randomized to receive ddI given either qd or bid in combination with d4T given bid (no doses specified).

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Documented HIV infection.
* CD4 cell count of at least 100 cells/mm3.
* Plasma HIV RNA count of 10,000 copies/ml or more within 14 days prior to study entry.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions and symptoms are excluded:

* Presence of a newly diagnosed AIDS-defining opportunistic infection requiring acute therapy at the time of enrollment.
* Bilateral peripheral neuropathy or signs and symptoms of bilateral peripheral neuropathy greater than or equal to Grade 2 at the time of screening.
* Inability to tolerate oral medication.
* Any other clinical condition that would preclude compliance with dosing requirements.

Patients with the following prior conditions are excluded:

* History of acute or chronic pancreatitis.
* Intractable diarrhea (6 or more loose stools/day for more than 7 consecutive days) within 30 days prior to study entry.
* Proven or suspected acute hepatitis within 30 days prior to study entry.

  1. Potent neurotoxic drugs, such as vincristine and thalidomide.
* Other anti-HIV therapy.

  1. Prophylaxis for pneumocystis carinii pneumonia (PCP) is strongly recommended for patients with CD4 cell counts less than or equal to 200/mm3 or who have had a prior episode of PCP.
* Immunizations recommended by ACIP for routine practice.
* Erythropoietin and G-CSF are allowed if myelosuppression emerges on study.

  1. Any antiretroviral therapy.
* Agents with significant systemic myelosuppressive, neurotoxic, pancreatotoxic, hepatotoxic, or cytotoxic potential within 3 months of study entry.

  1. Any prior antiretroviral therapy.
* Agents with significant systemic myelosuppressive, neurotoxic, pancreatotoxic, hepatotoxic, or cytotoxic potential within 3 months of study entry.

Active alcohol or substance abuse that would prevent adequate compliance or would increase the risk of pancreatitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-02; Primary Completion 2004-02 (Actual); Study Completion 2004-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Clinsites / Sorra Research Ctr, Birmingham, Alabama
  - Shared Med Research Foundation, Tarzana, California
  - Indiana Univ School of Medicine / Dept of Infect Dis, Indianapolis, Indiana
  - Medicine Faculty Associates, Ypsilanti, Michigan
  - New Jersey Community Research Initiative, Newark, New Jersey
  - ID Care Inc, Somerville, New Jersey
  - Fanno Creek Clinic, Portland, Oregon
  - Anderson Clinical Research, Pittsburgh, Pennsylvania
  - Univ of Texas Southwestern Med Ctr of Dallas, Dallas, Texas
  - Univ of Texas Med Branch, Galveston, Texas
  - Houston Clinical Research Network, Houston, Texas
  - Hampton Roads Med Specialists, Hampton, Virginia
  - Dr Iraj Mirshahi, Richmond, Virginia

REFERENCES:
- [Background] Mobley JE, Pollard RB, Schrader S, Adler MH, Kelleher T, McLaren C. Virological and immunological responses to once-daily dosing of didanosine in combination with stavudine. AI454-143 Team. AIDS. 1999 Jul 30;13(11):F87-93. doi: 10.1097/00002030-199907300-00003. PMID 10449279